CLINICAL TRIAL: NCT03547349
Title: The Effectiveness of the Jamboxx Respiratory Therapy Device in Treatment of Patients With Decreased Respiratory Function. Study 3: Post-Op Inpatients for Short Term Evaluation of Atelectasis
Brief Title: The Effectiveness of the Jamboxx Respiratory Therapy Device: Study 3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: My Music Machines Inc. (Industry)
Collaborators: Albany Medical College (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Jamboxx RT Device Study 3; 4R42HL132735-02 (NIH)
Record Dates: First submitted 2018-04-26; First posted 2018-06-06 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Atelectases, Postoperative Pulmonary
Keywords: respiratory therapy; videogaming therapy; incentive spirometry; atelectases
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Patients will be enrolled sequentially in Group 1 until the desired group enrollment number is met (N=25) at which point participants will be randomized into groups 2 and 3, stratified by surgery type (open or laproscopic)
Who Masked: Outcomes Assessor
Masking Description: Incidence and severity of atelectasis will be radiographically assessed on a 5 point scale (no apparent disease, subsegmental atelectasis, segmental atelectasis, lobar atelectasis, or pneumonia) by a chest radiologist and two pulmonary physicians blinded to study group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Group 1 (Active Comparator): These study patients will receive a study information/authorization sheet about the study prior to surgery during their pre-operative clinic visit. This subgroup will be provided postoperatively with a digital incentive spirometer connected to a tablet interface. This tablet device uses a digital interface to mimic the look and function of the standard issue incentive spirometer. Subjects in this group will receive current standard of care with routine surgical and RN encouragement to use the spirometer. The tablet will monitor and record spirometer device utilization.
  Interventions: Device: Digital Incentive Spirometer
- Group 2 (Active Comparator): These study patients will be consented by members of the research team prior to surgery at their pre-operative clinic visit. The patient will receive RT or RN education preoperatively as to the importance of incentive spirometry in prevention of post-operative respiratory complications. This subgroup will be provided with a digital incentive spirometer connected to a tablet interface. This tablet device uses a digital interface to mimic the look and function of the standard issue incentive spirometer, and will set a spirometry goal while collecting usage and pulmonary function data. Subjects in this group will also receive daily intensive education from a study team member during the postoperative time up until 72 hours or until discharge.
  Interventions: Device: Digital Incentive Spirometer
- Group 3 (Experimental): These study patients will be consented by a member of the research team prior to surgery at their pre-operative clinic visit. The patients will receive RT or RN education preoperatively as to the importance of incentive spirometry in prevention of post-operative respiratory complications. This subgroup will be provided with both intensive education reinforcement and the Jamboxx Respiratory Therapy Device that also includes multiple gaming programs. The games are meant to encourage incentive spirometry and are programmed to progress in accordance with the patient's personal increasing capacity. Subjects in this group will also receive daily intensive education from a study team member during the postoperative time up until 72 hours or until discharge.
  Interventions: Device: Digital Incentive Spirometer; Device: Jamboxx Respiratory Therapy Device

INTERVENTIONS:
Device: Digital Incentive Spirometer — This device is an incentive spirometer connected to a tablet interface. This tablet device uses a digital interface to mimic the look and function of the standard issue incentive spirometer
Device: Jamboxx Respiratory Therapy Device — THe Jamboxx Respiratory Therapy Device is a novel device that uses interactive gaming to encourage patient compliance with their prescribed respiratory therapy routines. The device consists of a computer game controller with mouthpiece, and breath flow sensor that connects to a tablet. With the Jamboxx Respiratory Therapy Device, users can choose from a suite of breath controlled respiratory therapy games to guide them through their routines while receiving real-time feedback, and long-term progress tracking.
  Arms: Group 3

SUMMARY:
The Effectiveness of the Jamboxx Respiratory Therapy Device in Treatment of Patients with Decreased Respiratory Function is a proposal for investigation of the application of gaming to improving respiratory health. The Jamboxx device (see appendix A for device details) combines gaming with traditional incentive spirometry to provide users with a fun experience to keep them engaged in their respiratory therapy routine. The device allows users to play a series of mini-games that walk them through their routines. The Jamboxx also records airflow and lung parameters with an external mouthpiece attachment to provide users with real time feedback, and helps to assess increases or decreases in relative lung function over time. The Jamboxx has the potential to significantly impact the field of respiratory therapy by being one of the first gaming devices for patient therapy, and the first respiratory therapy gaming device that is accessible to users with limited mobility. Jamboxx provides a fun and engaging, low cost alternative to the traditional therapy techniques used and aims to improve patient compliance.

This study addresses postoperative pulmonary atelectasis that results from diaphragm dysfunction and pain following upper abdominal surgery. This issue is a major cause of morbidity in these patients (Ford et al 1983). Incentive spirometry is used in this setting, but there is conflicting data regarding its effectiveness (Rupp et al 2013). Study 3 will focus on the questions regarding the influence of education and a novel use of a gaming device on prevention of atelectasis. Study 3 will include 3 subgroups of subjects. The first subject group will be enrolled in a nonintrusive observation only studies. Group 1 will explore the effect of technology via a tablet device on standard spirometry usage. Group 2 will look at the combined effect of technology via the tablet device and intensive education on compliance and reduction of post-surgical atelectasis. Finally, Group 3 will explore the effect of gaming technology with intensive educational reinforcement on compliance and reduction of post-surgical atelectasis.

DETAILED DESCRIPTION:
Testing Plan: Study participants will be enrolled sequentially in one of three study groups:

• Group 1 - the first 25 patients will be consented to participate by a member of the research team. These study patients will receive a study information/authorization sheet about the study prior to surgery during their pre-operative clinic visit. This subgroup will be provided postoperatively with an incentive spirometer connected to a tablet interface. This tablet device uses a digital interface to mimic the look and function of the standard issue incentive spirometer. Subjects in this group will receive current standard of care with routine surgical and RN encouragement to use the spirometer. The tablet will monitor and record spirometer device utilization. Demographic data (age ( or >89), gender, ethnicity) and body mass index (BMI) will be collected. No patient identifiers will be collected. At 72 hours or at discharge, the devices will be exchanged for standard issue incentive spirometer. Research staff will extract the demographic data described above as well as BMI.

Randomized Study Subgroups:

• Groups 2 and 3 are active study groups. -Patients will be randomized via a random number generator post-operatively to group 2 or 3, stratified by surgery type (laparoscopic or open) . Each subgroup will include a total of 72 randomized participants

Group 2 : These study patients will be consented by members of the research team prior to surgery at their pre-operative clinic visit. The patient will receive RT or RN education preoperatively as to the importance of incentive spirometry in prevention of post-operative respiratory complications. This subgroup will be provided with an incentive spirometer connected to a tablet interface. This tablet device uses a digital interface to mimic the look and function of the standard issue incentive spirometer, and will set a spirometry goal while collecting usage and pulmonary function data. Subjects in this group will also receive daily intensive education from a study team member during the postoperative time up until 72 hours or until discharge. This education will be done to reinforce the standard instruction provided by the hospital staff.

Research staff will collect data on pain, utilization of incentive spirometry, and room air oximetry. The oximetry measurements will be collected after patients have been off of oxygen for between 3.5 to 4 minutes. For patients requiring high levels of supplemental oxygen (pulse oximetry measurement (<90%), oxygen will not be removed for pulse oximetry measurements. The additional education and oximetry measure will be collected by a respiratory therapist three times a day at the preferred times of 0600, 1200 and 1800 post operatively. Patients will remain on study for 72 hours post-surgery, return to the OR, SICU admission or medical prescription of directed chest physiotherapy.

A Chest x-ray will be obtained at 48 hours post-surgery. Demographic data (age ( or >89), gender, ethnicity), pulmonary function data and body mass index (BMI) will be collected. No patient identifiers will be collected. At 72 hours or at discharge, the devices will be exchanged for standard issue incentive spirometer.

Group 3: These study patients will be consented by a member of the research team prior to surgery at their pre-operative clinic visit. The patients will receive RT or RN education preoperatively as to the importance of incentive spirometry in prevention of post-operative respiratory complications. This subgroup will be provided with both intensive education reinforcement and a spirometry tablet device that also includes multiple gaming programs. The games are meant to encourage incentive spirometry and are programmed to progress in accordance with the patient's personal increasing capacity.

This tablet device uses a digital interface to mimic the look and function of the standard issue incentive spirometer, and will set a spirometry goal while collecting usage and pulmonary function data. Subjects in this group will also receive daily intensive education from a study team member during the postoperative time up until 72 hours or until discharge. This education will be done to reinforce the standard instruction provided by the hospital staff.

Research staff will collect data on pain, utilization of incentive spirometry, and room air oximetry. The oximetry measurements will be collected after patients have been off of oxygen for between 3.5 to 4 minutes. For patients requiring high levels of supplemental oxygen (pulse oximetry measurement <90%),oxygen will not be removed for pulse oximetry measurements. The additional education and oximetry measure will be collected by a respiratory therapist three times a day at the preferred times of 0600, 1200 and 1800 post operatively. Patients will remain on study for 72 hours post-surgery, return to the OR, SICU admission or medical prescription of directed chest physiotherapy.

A Chest x-ray will be obtained at 48 hours post-surgery. Demographic data (age ( or >89), gender, ethnicity), pulmonary function data and body mass index (BMI) will be collected. No patient identifiers will be collected. At 72 hours or at discharge, the devices will be exchanged for standard issue incentive spirometer.

ELIGIBILITY:
Inclusion Criteria:

* Post-op patients with elective upper abdominal surgery including but not limited to: bariatric surgery, cholecystectomy, and bowel surgery

Exclusion Criteria:

* Patients who go directly to the ICU from the PACU post-surgery.
* Patients with visual impairments that make it difficult to understand written instructions
* Patients with hearing impairments that make it difficult to understand verbal instructions
* Patients who already receive supplemental oxygen therapy at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Severity of atelectasis | 48 hours post-surgery
  Severity of atelectasis radiographically assessed on a 5 point scale (1. no apparent disease, 2. subsegmental atelectasis, 3. segmental atelectasis, 4. lobar atelectasis, or 5. pneumonia) by a chest radiologist and two pulmonary physicians blinded to study group assignment. Within this scale range, no apparent disease represents the best possible outcome, while pneumonia represents the worst possible outcome

SECONDARY OUTCOMES:
Device Utilization Time | 72 hours post surgery or time of discharge, whichever comes first
  total usage time (in minutes) as recorded by the digital device
Device Uses | 72 hours post surgery or time of discharge, whichever comes first
  Total number of uses as recorded by the digital device
Pulse Oximetry | 3x/ day (except between hours of 10pm and 6am) until 72 hour post-surgery mark or time of discharge, whichever comes first
  Pulse Oximetry off of supplemental oxygen
Clinically relevant events | 72 hours post surgery or time of discharge, whichever comes first
  e.g. patient being sent for a chest x-ray, being ordered chest physiotherapy or increased oxygen requirement
Incidence of hospital acquired respiratory infection | 72 hours post surgery or time of discharge, whichever comes first
  Incidence of hospital acquired respiratory infection

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Fisher, MD, Study Chair — Albany Medical Center IRB
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No